CLINICAL TRIAL: NCT03164382
Title: A Phase III Randomized Trial of Comparison of Survival Benefit of Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil/Leucovorin With Sorafenib for Patients With Barcelona-Clinic Liver Cancer (BCLC)-C Stage Hepatocellular Carcinoma
Brief Title: Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil/Leucovorin Versus Sorafenib in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Zhao, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SB5010-2017-015
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Liver Cancer; Hepatic Carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Folfox protocol; Sorafenib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIF group (Experimental): FOLFOX regimen: oxaliplatin 130 mg/m2 on day 1 from hour 0 to 3; leucovorin 200 mg/m2 from hour 3 to 5, fluorouracil 400 mg/m2 bolus at hour 5, and then fluorouracil 2,400 mg/m2 over 46 hours, via hepatic artery, once every 3 weeks.
  Interventions: Drug: FOLFOX regimen
- Sorafenib group (Active Comparator): Sorafenib 200mg Tab, 400 mg twice per day orally. Treatment was given in 4-week cycles.
  Interventions: Drug: Sorafenib 200Mg Tab

INTERVENTIONS:
Drug: FOLFOX regimen — Firstly, the femoral artery was percutaneously punctured using the Seldinger technique. Then, the catheter was inserted into the celiac trunk or superior mesenteric artery for arteriography. When more than one feeding artery of HCC was detected, the smaller arteries were embolized with gelatin sponge particles. A micro-catheter was inserted through the arterial catheter located at the common hepatic artery or proper hepatic arterial branch (feeding artery). When blood flows into the gastroduodenal artery was confirmed by micro-catheter angiography, the route was embolized with a coil or micro-coil to prevent reflux of chemotherapeutic drugs to the stomach and duodenum. The peripheral part of the catheter that was exposed to the outside of the body was covered with medical sterile gauze and fastened on the thigh's skin using medical rubberized fabric and bandage. Catheter insertion was repeatedly performed before every cycle of treatment.
  Arms: HAIF group
Drug: Sorafenib 200Mg Tab — Sorafenib will be administered orally at the starting dose of 400 mg twice daily (800 mg total daily dose) to patients randomized to Arm S in accordance to its package insert or equivalent documentation. The 400 mg dose will be achieved by administration of 2 x 200 mg film-coated tablets, administered twice daily.
  Arms: Sorafenib group

SUMMARY:
This trial was designed to investigate whether the survival outcome, response rate and safety of hepatic arterial infusion of oxaliplatin, fluorouracil/leucovorin regimens for patients with Barcelona-Clinic Liver Cancer (BCLC)-C stage hepatocellular carcinoma was superior than those of the standard treatment with sorafenib or not.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is the fifth most common malignancy worldwide. Advanced-stage disease is found in 25%-70% of HCC at diagnosis, with a median survival time of only 4.2-7.9 months due to limited treatment options. To date, sorafenib is the only standard treatment shown to extend overall survival for advanced hepatocellular carcinoma (Ad-HCC). However, low response rates, modest survival advantages and high-level heterogeneity of individual response, such limitations of sorafenib prohibit its widespread use in Ad-HCC and more alternative therapies are highly required at present.

Hepatic arterial infusion chemotherapy (HAIC) can provide chemotherapeutic agents to liver at higher concentration with lower toxicity and has been reported favorable results in advanced HCC. However, HAIC provides good but variable outcomes, with a response rate of 7-81% and median survival time of 6-15.9 months. The unstable response may attribute to complicate combinations based on various drugs, including fluorouracil (5-FU), cisplatin, doxorubicin, mitomycin, leucovorin and interferon. FOLFOX (oxaliplatin, 5-FU/leucovorin) was a regimen first used in colon cancer with liver metastasis and reported to be effective both by systemic and HAIC in amounts of clinical trials. A recent phase II study has shown that HAI of FOLFOX (HAIF) was well tolerated and effective in Ad-HCC. To the investigator's knowledge, no clinical studies have been developed on comparing the survival benefit of HAIF with sorafenib for patients with Ad-HCC. In this phase III trial, the investigators aimed to compare survival outcome, response rate and safety of HAIF with sorafenib in patients with Ad-HCC.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any screening procedures.
* Cytohistological confirmation is required for diagnosis of HCC.
* Patients with advanced (unresectable and/or metastatic, stage C based on Barcelona-Clinic Liver Cancer [BCLC] staging classification) hepatocellular carcinoma which would not be suitable for treatment with loco-regional therapies or have progressed following locoregional therapy such as surgical resection, percutaneous hepatic arterial embolization, radiofrequency ablation, and percutaneous interventional therapy.
* At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1. Lesions previously treated with local therapy, such as radiation therapy, hepatic arterial embolization, radiofrequency ablation, and percutaneous interventional therapy should not be selected unless progression is noted at baseline, in which case, these lesions would be considered as non-target lesions.
* Current cirrhotic status of Child-Pugh class A-B, with no encephalopathy. Ascites controlled by diuretics is permitted in this study.
* Availability of a representative tumor tissue specimen (archival tumor tissue is allowed) at pre-screening.
* Eastern Cooperative Oncology Group Scale for Assessment of Patient Performance Status ≤ 2.
* Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and 4 weeks after the completion of trial.
* Adequate bone marrow, liver and renal function as assessed by central lab by means of the following laboratory requirements from samples within 7 days prior to procedure:

  * Hemoglobin > 100g/L
  * Absolute neutrophil count >3.0 ×109/L
  * Neutrophil count > 1.5 ×109/L
  * Platelet count ≥ 50.0 ×109/L
  * Total bilirubin < 51 μmol/L
  * Alanine transaminase (ALT) and aminotransferase (AST) < 5 x upper limit of normal
  * Albumin > 28 g/L
  * Prothrombin time (PT)-international normalized ratio (INR) < 2.3, or PT < 6 seconds above control
  * Serum creatinine < 110 μmol/L
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

* Received any prior systemic chemotherapy or molecular-targeted therapy for HCC such as sorafenib.
* Previous local therapy completed less than 4 weeks prior to the dosing and, if present any related acute toxicity > grade 1.
* Any contraindications for hepatic arterial infusion procedure:

  * Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).
  * Renal failure / insufficiency requiring hemo-or peritoneal dialysis.
  * Known severe atheromatosis.
  * Known uncontrolled blood hypertension (> 160/100 mm/Hg).
* Patients with any other malignancies within the last 3 years before study start.
* History of HCC tumor rupture.
* Patients with severe encephalopathy.
* Patients with known active bleeding (e.g. from GI ulcers, esophageal varices) within 2 months prior to baseline/screening visit or with history or evidence of inherited bleeding diathesis or coagulopathy.
* Clinically significant (CTC grade 3 or 4) venous or arterial thrombotic disease within past 6 months.
* History of cardiac disease:

  * Congestive heart failure >New York Heart Association (NYHA) class 2 (refer to Appendix 13.9).
  * Active coronary artery disease (CAD) (myocardial infarction more than 6 months prior to study entry is allowed).
  * Cardiac arrhythmias (>Grade 2 NCI-CTCAE Version 4.0) which are poorly controlled with anti-arrhythmic therapy or requiring pace maker.
  * Uncontrolled blood hypertension (> 160/100 mm/Hg).
* Serious, non-healing wound, ulcer, or bone fracture.
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within past 6 months prior to study treatment.
* Clinically significant third space fluid accumulation (i.e., ascites requiring tapping despite use of diuretic or pleural effusion that either required tapping or is associated with shortness of breath).
* Patients who have undergone major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks of the start of protocol treatment.
* History of a bone marrow or solid organ transplant.
* Use of biologic response modifiers, such as G-colony stimulating factor (CSF), within 3 weeks prior to start of study drug. (G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however, they may not be substituted for a required dose reduction). Subjects taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 1 month prior to the study or during the study.
* Any other condition that would, in the Investigator's judgment, contraindicate patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable or unwilling to swallow medication, social/ psychological issues, etc.
* Unable to undergo either contrast-enhanced magnetic resonance imaging (MRI) or contrast-enhanced computed tomography (CT).
* Known history of human immunodeficiency virus (HIV) seropositivity. HIV testing is not required as part of this study.
* Patients who have received any other investigational agents within a period of time that is less than the cycle length used for that treatment or equal to 4 weeks (whichever is shorter) prior to starting study drug and recovered from any side effects to grade 1 or less.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 7 days after permanently discontinuing HAIF and/or sorafenib treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
  * Combination of any two of the following (a+b or a+c, or b+c):

    1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    2. Placement of an intrauterine device or intrauterine system
    3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

* Sexually active males unless they use a condom during intercourse while receiving treatment and for 7 days after stopping study treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Subjects unable to suffer the discomfort of the HAI procedure (e.g. pain, claustrophobia, noise).
* Any contraindication for sorafenib, oxaliplatin, leucovorin, or fluorouracil administration.
* Any agents which could affect the absorption or pharmacokinetics of the study drugs.
* Known or suspected allergy to the investigational agents or any agent given in association with this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 months
  Overall survival was the length of time after treatment until death from any cause.

SECONDARY OUTCOMES:
Time to Progression | 1 months
  Time to Progression was defined as the time from commencement of treatment to radiological disease progression.
Time to Intrahepatic tumor Progression | 1 months
  Time to Intrahepatic tumor Progression was defined as the time from commencement of treatment to radiological intrahepatic tumor progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Minimally Invasive Interventional Division, Department of Medical Imaging and Interventional Radiology, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen QF, Jiang X, Hu Y, Chen S, Lyu N, Zhao M. Interventional arterial chemotherapy versus sorafenib for advanced hepatocellular carcinoma in China: a health economic evaluation of open-label, randomised, phase 3 study. BMJ Open. 2025 May 27;15(5):e095508. doi: 10.1136/bmjopen-2024-095508. PMID 40436447
- [Derived] Lyu N, Wang X, Li JB, Lai JF, Chen QF, Li SL, Deng HJ, He M, Mu LW, Zhao M. Arterial Chemotherapy of Oxaliplatin Plus Fluorouracil Versus Sorafenib in Advanced Hepatocellular Carcinoma: A Biomolecular Exploratory, Randomized, Phase III Trial (FOHAIC-1). J Clin Oncol. 2022 Feb 10;40(5):468-480. doi: 10.1200/JCO.21.01963. Epub 2021 Dec 14. PMID 34905388